CLINICAL TRIAL: NCT02741336
Title: Electrophysiologic Changes in Blacks Treated With CBT for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Daniel Cukor, Principle Investigator, National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Organization: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 675013
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Blood Glucose Self-Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-I Intervention (Experimental): For those randomized to the CBT-I group, the therapist will initiate telephone-delivered cognitive-behavioral therapy within 2 weeks of baseline assessment. Participants will complete 4 telephone sessions over a period of 8 weeks. Sessions last approximately 45 minutes. CBT-I is a short-term, focused psychotherapy that is action-oriented, practical, rational, and helps the patient gain independence and effectiveness in dealing with real-life issues. Techniques utilized in CBT-I include psychoeducation, sleep hygiene, cognitive restructuring, stimulus control, sleep restriction, and relaxation training.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
- Self-Monitoring Control Group (Active Comparator): Individuals randomized to the self-monitoring control group will be asked to complete a weeklong sleep diary every other week for 8 weeks. The sleep diary will inquire about (1) the time of getting into bed; (2) the time at which the individual attempted to fall asleep; (3) sleep onset latency; (4) number of awakenings; (5) duration of awakenings; (6) time of final awakening; (7) final rise time; (8) perceived sleep quality (rated via Likert scale); and (9) an additional space for open-ended comments from the respondent. The control condition is designed to increase self-monitoring, which has been demonstrated to be an effective means of inducing change for various health behaviors such as diet and exercise.
  Interventions: Behavioral: Self-Monitoring

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — Cognitive-behavioral therapy is a short-term, focused psychotherapy for a wide range of psychological and behavioral issues including depression, anxiety, anger, and non-compliance. The focus of the intervention is on how one thinks, behaves, and communicates in real time, as opposed to a focus on one's early childhood experiences. The therapist assists the patient in identifying specific distortions and biases in thinking and provides guidance on how to modify these beliefs. CBT helps the patient learn effective self-help skills that are used in homework assignments that ultimately help change the way one thinks, feels and behaves. The
  ￼ intervention is action-oriented, practical, rational, and helps the patient gain independence and effectiveness in dealing with real-life issues. Techniques utilized in CBT-I include psychoeducation, sleep hygiene, cognitive restructuring, stimulus control, sleep restriction, and relaxation training.
  Arms: CBT-I Intervention
Behavioral: Self-Monitoring
  Arms: Self-Monitoring Control Group

SUMMARY:
Insomnia is a highly prevalent, often debilitating, and economically burdensome condition. Reviews of the literature indicate that there are ethnic differences in sleep behavior, with African Americans objectively and subjectively reporting more disordered sleep than Caucasian Americans.Chronic insomnia can have a significant impact on mental and physical health outcomes and has been associated with impaired cognitive performance, particularly, in areas of speed, attention, working memory, and executive function. In order to understand the brain mechanisms in sleep disorder both during resting state as well as during cognitive processing, the investigators will assess resting state EEG (during eyes-closed and eyes-open conditions) as well as ERP tasks for assessing decision-making and reward processing. The primary objective of the study is to evaluate the effect of a tailored, telephone-delivered cognitive behavioral intervention, versus a self- monitoring control condition, on symptoms of insomnia and its neurodynamic correlates.

Hypotheses: Among Blacks subjectively reporting symptoms of insomnia, those randomized to the tailored, telephone-delivered CBT-I, compared with those randomized to the self-monitoring control group, will have: Hyp. 1: Greater reduction in symptoms of insomnia as measured by the Pittsburgh Sleep Quality Index. Hyp. 2: Greater neurophysiologic improvement (ERP, ERO) in the intervention condition in response to laboratory paradigms Hyp 3: Greater improvement in psychosocial functioning including reduction in depression and increase in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* A positive endorsement of insomnia items on the Sleep Disorders Questionnaire
* Self- reported race/ethnicity as black (men and women)
* Ages 30 to 50 years
* Accessible by telephone
* No plans to move away from the region within the year following enrollment
* Consent to participate.

Exclusion Criteria:

* Documented co-existing sleep apnea
* Self-reported use of sleep medication
* Impaired cognitive or functional ability precluding meaningful participation
* Stated intention to move within the same year of enrollment.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Sleep Diary | 2 months after enrollment

SECONDARY OUTCOMES:
QEEG tests of cognition | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States